CLINICAL TRIAL: NCT01323543
Title: "Elaspine™ Implant System Post Marketing Clinical Study: A Prospective, Multicentre Study to Evaluate the Safety and Performance of the Elaspine™ System in the Surgical Treatment of Degenerative Lumbar Spine"
Brief Title: Safety and Performance of the Elaspine System in the Treatment of the Lumbar Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinelab AG (Industry)
Collaborators: UL International GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10k002 PMCS 01
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Lower Back Pain
Keywords: Back Pain,; Back Pains, Low; Low Back Pains; Pain, Low Back; Pains, Low Back; Lumbago; Lower Back Pain; Back Pain, Lower; Back Pains, Lower; Lower Back Pains; Pain, Lower Back; Pains, Lower Back; Low Back Ache; Ache, Low Back; Aches, Low Back; Back Ache, Low; Back Aches, Low; Low Back Aches; Low Backache; Backache, Low; Backaches, Low; Low Backaches; Low Back Pain, Recurrent; Recurrent Low Back Pain; Low Back Pain, Postural; Postural Low Back Pain; Low Back Pain, Mechanical; Mechanical Low Back Pain; Low Back Pain, Posterior Compartment
MeSH Terms: conditions — Low Back Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elaspine™ (Experimental): Impantation of Elaspine™ device
  Interventions: Device: Elaspine™

INTERVENTIONS:
Device: Elaspine™ — Implantation of device

SUMMARY:
The safety and performance of the Elaspine™ Implant System in the treatment of lower back pain will be evaluated with a prospective and nonrandomized, multicenter post-marketing clinical study (PMCS). The study will be enrolled within Germany and Switzerland in 3-5 clinical centres, including in average 10 patients per centre. The study is conducted in accordance with the Standard ISO 14155, where applicable on clinical investigation of medical devices for human subjects and other legal requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed and understood the approved Informed Consent form and is able to meet the proposed follow-up and postoperative management program.
2. Patient is skeletally mature and between 21 - 80 years of age.
3. Patient's pre-operative Body Mass Index (BMI) is ≤ 34.
4. Patient's pre-operative Oswestry Disability Index (ODI) is ≥ 30% (≥15 out of 50 points).
5. Patient's pre-operative back pain Visual Analogue Scale (VAS) is >60 (0-100 scale), with or without associated leg pain (leg pain VAS score).
6. Patient has received non-operative treatment for low back pain for > 6 months and is unresponsive.
7. Patient has one or more of the following structural abnormalities with imaging studies verifying them at one or two contiguous levels within L1-L5:

   * Discopathy
   * Degenerative disc disease
   * Massive or recurrent disc herniation
   * Non-isthmic spondylolisthesis ≤ Grade 1 (acc. To Meyerding)
   * Spinal stenosis
   * Partially defective facet joints
   * Retrolisthesis according to one of the following definitions (acc. to Ruch, William J.; Literature Reference 21):

     * Complete Retrolisthesis: The body of one vertebra is posterior to both the vertebral body of the segment of the spine above as well as below
     * Stairstepped Retrolisthesis: The body of one vertebra is posterior to the body of the spinal segment above, but is anterior to the one below.
     * Partial Retrolisthesis: The body of one vertebra is posterior to the body of the spinal segment either above or below.

Exclusion Criteria:

1. Degenerative spondylolisthesis greater than Grade 1 as defined by greater than 25 percent vertebral slip forward over the inferior vertebral body (acc. to Meyerding Classification) or significant segmental instability at or adjacent to intended treatment level.
2. Need for more than two-level or two non-contiguous-level surgery in the lumbar spine.
3. Patient has more than 50% defective facet joint (half of the articular joint surface) or laminectomy
4. Patient is scheduled for another lumbar surgery such as but not limited to a fusion
5. Patient has recent vertebral fractures or past fractures which did not heal.
6. Patient has known allergies to titanium alloy and polycarbonate urethane (PCU).
7. Patient has clinically compromised vertebral body structure and morphology at the lumbar spine due to current or past trauma (or pathological vertebral fracture) or significant endplate incompetence such as Schmorl´s node.
8. Patient has spondylolysis at the levels to be treated or an adjacent level.
9. Patient has a frontal curve in the lumbar spine >10°.
10. Patient has previously been diagnosed osteopenia or metabolic bone diseases or severe osteoporosis - if suspected to be confirmed by bone density being 2.5 SD below normal as assessed using DEXA analysis in:

    * Postmenopausal females if suggested by x-ray or other risk factors
    * Males over the age of 60 that have sustained a non-traumatic hip or spine fracture
11. Patient is taking medications known to potentially interfere with bone/soft tissue healing, including but not limited to the long term use of corticosteroids. (This is not intended to exclude patients using inhalation medications for asthma.)
12. Patient has an active infection either systemic or at the local site of intended surgery.
13. Patient has been diagnosed with hepatitis, rheumatoid arthritis, an autoimmune disease, or AIDS, ARC, or is HIV positive or any other diseases that according to surgeons may have an impact on the outcome of the surgery.
14. Patients with known malignant diseases or bone tumors.
15. Patients with vascular malformations such as abdominal aneurysm.
16. Patient has a progressive neuromuscular disease. Patient has active malignancy within the last 15 years, unless the malignancy was treated with curative intent and there have been no clinical signs or symptoms for at least 5 years.
17. Patient has cervical myelopathy.
18. Patient is pregnant or planning in becoming pregnant in the next 2 years.
19. Patient is currently participating in another investigational study where the endpoints have not yet been achieved. 8/35 Elaspine™ PMCS 01, Clinical Investigation Plan CIP EN Version C, October 1st, 2010 CONFIDENTIAL
20. Patient has mental illness, and/or diagnosed as clinically depressed or belongs to a vulnerable population (e.g., prisoner, severe drug abuser, developmentally disabled) that would compromise ability to provide informed consent or compliance with follow-up requirements. If suspected to be confirmed by classification according to DSM IV.
21. Patient has had another surgical procedure(s) within the last 60 days involving general anesthesia or any surgical procedure that might increase the risk of deep vein thrombosis.
22. Loss of Disk height according to Pfirrmann (> C) or Frymoyer (>3) and or severe spondylosis.
23. Patient shows three or more signs of anorganic behaviour (Waddell´s signs).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Safety | 24 months
  Incidence (including severity) of operative and post-operative complications throughout the first 3 months postoperatively by category (general, operative, post-operative, possibly device related etc.)
Performance | 24 months
  Defined as the incidence of device complications and device malfunctions (including severity), as assessed by radiographic evaluation throughout the first 12 months post-operatively. Device malfunctions include, but are not limited to loosening or breakage of the pedicle screws, disassembly of the locking clip, breakage of the rod, pathological motion or stiffness of the segments and disc collapse. Reading of the imaging studies will be centralized at an independent facility.

SECONDARY OUTCOMES:
Changes in function status (ODI), back pain (VAS) and health status (SF-12) at two-years post-operatively will be measured and compared to the preoperative baseline | 24 months
Changes in neurologic function at two-years post-operatively as compared to the preoperative baseline by motor, sensory, reflexes and straight leg raise | 24 months
Changes in angular range of motion from maximum flexion to extension between preoperative baseline and the two-year postoperative outcome assessed by radiographic imaging (dynamic xrays) | 24 months

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (4):
  - Helios Rosmann Klinik, Breisach, Baden-Wurttemberg
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - HSK Dr. Horst-Schmidt-Klinik, Wiesbaden, Hessia
  - Katholisches Klinikum Marienhof, Koblenz, Rhineland-Palatinate
- HUG Hôpitaux Universitaires de Genève, Geneva, Canton of Geneva, Switzerland